CLINICAL TRIAL: NCT01897493
Title: Effect of Evacetrapib on the Pharmacokinetics of Digoxin in Healthy Subjects
Brief Title: A Study of Evacetrapib and Digoxin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14619; I1V-MC-EIAQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — evacetrapib; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Digoxin (Active Comparator): 0.5 milligram (mg) digoxin administered orally once daily (QD) on Day 1
  Interventions: Drug: Digoxin
- Evacetrapib + Digoxin (Experimental): 130 mg evacetrapib administered orally, QD for 14 days (Days 6 through 19) with a single oral dose of 0.5 mg digoxin coadministered on Day 15
  Interventions: Drug: Evacetrapib; Drug: Digoxin

INTERVENTIONS:
Drug: Evacetrapib — Administered orally
  Other Names: LY2484595
  Arms: Evacetrapib + Digoxin
Drug: Digoxin — Administered orally

SUMMARY:
The main purpose of this study is to determine how much digoxin gets into the blood stream and how long it takes the body to get rid of it when given with the study drug evacetrapib. This study will also look at the effect of evacetrapib on the removal of digoxin from the body by the kidneys. Information about any side effects that may occur will be collected. This study will last approximately 33 days for each participant, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males and females (of non-childbearing potential)
* Have a body mass index of 18 to 32 kilograms per square meter (kg/m^2)
* Normal renal function

Exclusion Criteria:

* Participants who currently smoke or use tobacco or nicotine products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Evacetrapib+Digoxin: Period 1 (Day 1 through Day 6 predose): Participants received a single oral dose of 0.5 milligrams (mg) digoxin on Day 1 Period 2 (Day 6 postdose through Day 20): Participants received an oral dose of 130 mg evacetrapib once daily (QD) on Days 6 through 19 with single oral dose of 0.5 mg digoxin administered on Day 15
Period: Period 1 (Day 1 Through Day 6 Predose)
Arm/Group | Evacetrapib+Digoxin
Started | 16
Received at Least 1 Dose of Study Drug | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Period 2 (Day 6 Postdose Through Day 20)
Arm/Group | Evacetrapib+Digoxin
Started | 15
Received at Least 1 Dose of Study Drug | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Evacetrapib+Digoxin: Period 1 (Day 1 through Day 6 Predose): Participants received a single oral dose of 0.5 mg digoxin on Day 1 Period 2 (Day 6 Post-Dose through Day 20): Participants received an oral dose of 130 mg evacetrapib QD on Days 6 through 19 with a single oral dose of 0.5 mg digoxin administered on Day 15
Arm/Group | Evacetrapib+Digoxin
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Digoxin
Time Frame: Periods 1 and 2: digoxin predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours after administration of digoxin
Population: All enrolled participants who received digoxin in Periods 1 and 2 and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- Period 1-Digoxin: Digoxin: Participants received 0.5 mg digoxin administered orally QD on Day 1
- Period 2-Evacetrapib + Digoxin: Evacetrapib+Digoxin: Participants received 130 mg evacetrapib administered orally, QD for 14 days (Days 6 through 19) with a single oral dose of 0.5 mg digoxin coadministered on Day 15
Arm/Group | Period 1-Digoxin | Period 2-Evacetrapib + Digoxin
Number analyzed (Participants) | 16 | 15
nanograms/milliliter (ng/mL) | 1.75 (28) | 2.15 (32)

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC0-∞) of Digoxin
Time Frame: as for outcome 1
Population: All enrolled participants who received digoxin in Periods 1 and 2 and had evaluable AUC0-∞ data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | Period 1-Digoxin | Period 2-Evacetrapib + Digoxin
Number analyzed (Participants) | 16 | 15
nanograms*hour/milliliter (ng*h/mL) | 31.3 (18) | 33.5 (26)

3. Primary Outcome: PK: Time of Maximum Observed Drug Concentration (Tmax) of Digoxin
Time Frame: as for outcome 1
Population: All enrolled participants who received digoxin in Periods 1 and 2 and had evaluable tmax data.
Measure: Median (Full Range); unit: hours
Arm/Group | Period 1-Digoxin | Period 2-Evacetrapib + Digoxin
Number analyzed (Participants) | 16 | 15
hours | 2.00 [1.00 to 2.00] | 2.00 [1.00 to 2.00]

4. Secondary Outcome: Renal Clearance (CLr) of Digoxin
Description: CLr was defined as the volume of serum cleared of digoxin per unit of time after a single dose of digoxin.
Time Frame: as for outcome 1
Population: All enrolled participants who received digoxin in Periods 1 and 2 and had evaluable CLr data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/hour (L/h)
Arm/Group | Period 1-Digoxin | Period 2-Evacetrapib + Digoxin
Number analyzed (Participants) | 16 | 15
liters/hour (L/h) | 9.43 (14) | 8.10 (18)

ADVERSE EVENTS:
Groups:
- Digoxin: Digoxin: Participants received a single dose of 0.5 mg digoxin administered orally on Day 1. Adverse events (AEs) are reported through predose on Day 6
- Evacetrapib: Evacetrapib: Participants received 130 mg evacetrapib administered orally, alone, QD for Days 6 up to 15. AEs are reported from post-dose on Day 6 through predose of Digoxin on Day 15.
- Evacetrapib + Digoxin: Evacetrapib+Digoxin: Participants received 130 mg evacetrapib administered orally, QD for 14 days (Days 6 to 19) with a single oral dose of 0.5 mg digoxin coadministered on Day 15. AEs are reported from post-dose on Day 15 up to Day 33.
Arm/Group | Digoxin | Evacetrapib | Evacetrapib + Digoxin
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/16 | 1/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digoxin (N=16) | Evacetrapib (N=15) | Evacetrapib + Digoxin (N=15)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days